CLINICAL TRIAL: NCT01442376
Title: A Multicenter, Randomized, Double-blind, Parallel Group Study to Evaluate the Efficacy and Safety of Two Different Doses of Palonosetron Compared to Ondansetron in the Prevention of CINV in Pediatric Patients Undergoing Single and Repeated Cycles of MEC or HEC
Brief Title: Efficacy and Safety of Palonosetron Intravenous in Prevention of Chemotherapy Induced Nausea and Vomiting in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PALO-10-20
Record Dates: First submitted 2011-09-21; First posted 2011-09-28 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting
Keywords: Prevention of Chemotherapy-Induced Nausea and Vomiting; Palonosetron; Ondansetron; Pediatric
MeSH Terms: conditions — Vomiting | interventions — Palonosetron; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Palonosetron 10 mcg/kg (Experimental): Palonosetron and placebo to Ondansetron
  Intervention:
  Drug: Palonosetron
  Interventions: Drug: Palonosetron; Drug: Placebo to Ondansetron
- Palonosetron 20 mcg/kg (Experimental): Palonosetron and placebo to Ondansetron
  Intervention:
  Drug: Palonosetron
  Interventions: Drug: Palonosetron; Drug: Placebo to Ondansetron
- Ondansetron (Active Comparator): Ondansetron and placebo to Palonosetron
  Drug:
  Comparator: Ondansetron
  Interventions: Drug: Ondansetron; Drug: Placebo to Palonosetron

INTERVENTIONS:
Drug: Palonosetron — Single dose Palonosetron IV 10 mcg/kg up to a maximum total dose of 0.75 mg
  Arms: Palonosetron 10 mcg/kg
Drug: Palonosetron — Single dose Palonosetron IV 20 mcg/kg up to a maximum total dose of 1.5 mg
  Arms: Palonosetron 20 mcg/kg
Drug: Ondansetron — Single three (every 4 hours) Ondansetron IV doses 0.15 mg/kg up to a maximum total dose of 32 mg
  Arms: Ondansetron
Drug: Placebo to Ondansetron
  Arms: Palonosetron 10 mcg/kg
Drug: Placebo to Ondansetron
  Arms: Palonosetron 20 mcg/kg
Drug: Placebo to Palonosetron
  Arms: Ondansetron

SUMMARY:
The primary objective is to evaluate the efficacy of two different doses of IV palonosetron in the prevention of chemotherapy induced nausea and vomiting in MEC and HEC patients through 120 hours after start of chemotherapy in single and repeated chemotherapy cycles. The secondary objectives are to evaluate the safety and tolerability of IV palonosetron in pediatric patients and evaluate the pharmacokinetics of IV palonosetron in a subset of pediatric CINV patients.

DETAILED DESCRIPTION:
For neonates (<28 days, full term) an open-label sub-study will be conducted to assess exposure and tolerability in this age group with escalating doses of palonosetron, starting with 3 mcg/kg to the first three or more neonates included in the study. If this dose is shown to be safe and well tolerated then the following three neonates will be treated with a dose of 10 mcg/kg. If also this dose is safe and well tolerated, then the following three neonates will be treated with a dose of 20 mcg/kg. If this last dose is also shown to be safe and well tolerated, then all the following neonates will be randomized to the main study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed by parent(s)/legal guardians of the pediatric patient in compliance with the local laws and regulations. In addition signed children's assent form according to local requirements
* Male or female in- or out-patients from neonates (full term) to <17 years at the time of randomization
* Patient weight at least 3.2 kg
* Histologically, and/or cytologically (or imaging in the case of brain tumors) confirmed malignant disease
* Naïve or non-naïve to chemotherapy
* Scheduled and eligible to receive at least one of the moderately or highly emetogenic chemotherapeutic agents on Study Day 1
* For patients aged ≥ 10 years to <17 years: ECOG PS ≤ 2
* For patients with known hepatic impairment: in the Investigator's opinion the impairment should not jeopardize patient's safety during the study
* For patients with known renal impairment: in the Investigator's opinion the impairment should not jeopardize patient's safety during the study
* For patients with known history or predisposition to cardiac abnormalities: in the Investigator's opinion the history/predisposition should not jeopardize patient's safety during the study
* For patients with known clinically relevant abnormal laboratory values: in the Investigator's opinion the abnormality should not jeopardize the patient's safety during the study
* Fertile patients (male or female) must use reliable contraceptive measures
* Female patients who have attained menarche must have a negative pregnancy test at the screening visit (Visit 1) and at study treatment visit (Visit 2)

Exclusion Criteria:

* Lactating or pregnant female patient
* Patient has received total body irradiation, upper abdomen radiotherapy, radiotherapy of the cranium, craniospinal regions or the pelvis within 1 week prior to study entry (screening)
* Scheduled to receive concomitant total body irradiation, radiotherapy of the upper abdomen, lower thorax region, or cranium/craniospinal regions up to 24 hours after study drug administration
* Known history of allergy to any component or other contraindications to any 5-HT3 receptor antagonists
* Active infection
* Uncontrolled medical condition
* Marked baseline prolongation of QTc interval [QTcB or QTcF > 460 msec] in any of the ECG assessments at screening. For this purpose, assessment will rely on the automatic interpretation by the ECG machine
* Patient suffering from ongoing vomiting from any organic etiology (including patients with history of gastric outlet obstruction or intestinal obstruction due to adhesions or volvulus) or patients with hydrocephalus
* Patient who experienced any vomiting, retching, or nausea within 24 hours prior to the administration of the study drug
* Patient who received any drug with potential anti-emetic effect within 24 hours prior to administration of study treatment, including but not limited to:
* NK1- receptor antagonists (e.g. aprepitant)
* 5-HT3 antagonists (e.g., ondansetron, granisetron, dolasetron);
* Phenothiazines (e.g., perphenazine, prochlorperazine, promethazine, fluphenazine, chlorpromazine, thiethylperazine);
* Butyrophenones (e.g., droperidol, haloperidol);
* Benzamides (e.g., metoclopramide, alizapride);
* Corticosteroids (e.g., prednisone, methylprednisolone; except inhaled steroids for respiratory disorders and topical steroids for skin disease with doses of ≤ 10 mg of prednisone daily or its equivalent); Corticosteroids foreseen in the chemotherapy regimen or to reduce intracranial pressure are allowed. According to the guidelines1,2, patients will receive also dexamethasone as a co-medication in accordance with standard clinical practice and if deemed appropriate by the Investigator.
* Dimenhydrinate; Hydroxyzine; Domperidone; Lorazepam; Cyclizine; Cannabinoids; Scopolamine; Trimethobenzamide HCl; Meclizine hydrochloride; Pseudoephedrine HCl;
* Over the Counter (OTC) antiemetics, OTC cold or OTC allergy medications;
* Herbal preparations containing ephedra or ginger.
* Patient aged ≤ 6 years who received any investigational drug (defined as a medication with no marketing authorization granted for any age group and any indication) within 90 days prior to Day 1, or patient aged > 6 years who received any investigational drug within 30 days prior to Day 1 or is expected to receive investigational drugs prior to study completion
* Patient who participated in any previous trial with palonosetron

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 502 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (67):
- United States (14):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - The Children's Hospital, Aurora, Colorado
  - A. I. duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Nemours Children's Clinic, Pensacola, Florida
  - Backus Children's Hospital at University Pediatrics, Savannah, Georgia
  - University of Kentucky - Chandler Medical Center, Lexington, Kentucky
  - Upstate Medical University, Syracuse, New York
  - Department of Pediatrics, Valhalla, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Cook Children's Medical Center, Fort Worth, Texas
- Argentina (4):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - CEMIC, Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Hospital Nacional "Prof. Dr. Alejandro Posadas", El Palomar
- Austria (2):
  - Children's Cancer Research Institute, Vienna
  - Medical University of Vienna, Vienna
- Bulgaria (3):
  - Pediatrics and Genetic Medicine Clinic, Plovdiv
  - Specialised Hospital for Active Treatment of Oncohematological Diseases in Children, Sofia
  - Specialised Pediatric Clinic of Clinical Hematology and Oncology Mutiprofile Hospital for Active Treatment "Sveta Marina", Varna
- Chile (4):
  - Hospital Dr Luis Calvo Mackenna, Santiago
  - Clinica Santa Maria SA, Santiago
  - Hospital Clinico UC, Santiago
  - Clinica Davila, Santiago
- Czechia (4):
  - University Hospital Brno, Children's Medical Centre, Clinic of Pediatric Oncology, Brno
  - University Hospital in Ostrava, Clinic of Pediatric, Ostrava
  - University Hospital in Pilsen, Plzen-Lochotin
  - University Hospital Motol, Department of Paediatric Heamatology and Oncology, Prague
- Estonia (2):
  - Tallin Children's Hospital, Tallinn
  - Tartu University Hospital, Hematology - Oncology Clinic, Tartu
- France (3):
  - CHRU de Lille - Hopital d'Hematologie Pediatrique, Lille
  - Hopital Arnaud de Villenueve, Montpellier
  - CHRU de Tours - Centre de Pediatrie Gatien de Clocheville, Tours
- Germany (2):
  - University Hospital of Cologne, Cologne
  - University Medical Center Freiburg, Freiburg im Breisgau
- Hungary (2):
  - Semmelweis University, 2nd Department of Pediatrics, Budapest
  - University of Szeged, Szent-Gyorgyl Albert Clinical Center, Department of Pediatrics, Szeged
- Peru (3):
  - Instituto Nacional de Enfermedades Neoplásicas, Lima
  - Oncosalud SAC RCI 300, Lima
  - Clinica Anglo Americana - Centro de Investigacion Oncologica CAA, San Isidro Lima
- Poland (6):
  - Szpital Uniwersytecki - Department of Pediatrics, Hematology and Oncology, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Uniwersytecki Szpital, Lodz
  - Dzieciecy Szpital Kliniczny, Lublin
  - Institut Pomnik - The Children Memorial Health Institute, Department of Oncology, Warsaw
  - Samodzielny Publiczny Szpital, Wroclaw
- Romania (4):
  - Fundeni Clinical Institute, Pediatrics Clinic, Bucharest
  - "Prof. Dr. Alexandru Trestioreanu" Institute of Oncology, Pediatric Oncology Department, Bucharest
  - "Prof. Dr. Ion Chiricuta" Institute of Oncology, Cluj-Napoca Pediatric Department, Cluj-Napoca
  - Sf. Maria - Chidren's Emergency Clinical Hospital, Iași
- Russia (8):
  - Chelyabinsk Pediatric Regional Clinical Hospital, Oncohematology Department, Chelyabinsk
  - Pediatric Regional Clinical Hospital, Krasnodar
  - Russian Oncology Research Center, Moscow
  - Moscow State Institution: Morozovskaya Pediatric City Clinical Hospital, Moscow
  - Omsk Regional Clinical Oncology Center, Omsk
  - St. Petersburg State Medical University, Saint Petersburg
  - State Clinical Hospital, Saint Petersburg
  - Regional Pediatric Clinical Hospital #1, Yekaterinburg
- Serbia (2):
  - Department for hematology and oncology, Belgrade
  - Clinical Center Nis, Clinic for pediatrics internal diseases, Department for hematology and oncology, Niš
- Ukraine (4):
  - State Institution: V. K. Husak Institute of Urgent and Reconstructive Surgery, Donetsk
  - Public Treatment and Prophylaxis Institution: Regional Children's Clinical Hospital, Donetsk
  - Public Healthcare Institution: Regional Children's Clinical Hospital #1, Kharkiv
  - National Institute of Cancer, Kyiv

REFERENCES:
- [Derived] Kovacs G, Wachtel AE, Basharova EV, Spinelli T, Nicolas P, Kabickova E. Palonosetron versus ondansetron for prevention of chemotherapy-induced nausea and vomiting in paediatric patients with cancer receiving moderately or highly emetogenic chemotherapy: a randomised, phase 3, double-blind, double-dummy, non-inferiority study. Lancet Oncol. 2016 Mar;17(3):332-344. doi: 10.1016/S1470-2045(15)00520-3. Epub 2016 Jan 19. PMID 26795844

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 502 patients were enrolled and randomly assigned to treatment. Study drug was not administered to 8 randomized patients, of these patients 2 had also an adverse event and were counted under this category in overall study statement. Therefore 494 patients did receive the study drug and are part of the analysis for the safety population.
Groups:
- Palonosetron 10 mcg/kg: Palonosetron and placebo to Ondansetron
  Intervention:
  Drug: Palonosetron
  Palonosetron: Single dose Palonosetron IV 10 mcg/kg up to a maximum total dose of 0.75 mg
  Placebo to Ondansetron
- Palonosetron 20 mcg/kg: Palonosetron and placebo to Ondansetron
  Intervention:
  Drug: Palonosetron
  Palonosetron: Single dose Palonosetron IV 20 mcg/kg up to a maximum total dose of 1.5 mg
  Placebo to Ondansetron
- Ondansetron: Ondansetron and placebo to Palonosetron
  Drug:
  Comparator: Ondansetron
  Ondansetron: Single three (every 4 hours) Ondansetron IV doses 0.15 mg/kg up to a maximum total dose of 32 mg
  Placebo to Palonosetron
Period: Overall Study
Arm/Group | Palonosetron 10 mcg/kg | Palonosetron 20 mcg/kg | Ondansetron
Started | 169 (Randomized patients) | 169 (Randomized patients) | 164 (Randomized patients)
Completed | 166 | 160 | 159
Not Completed | 3 | 9 | 5
Not completed — Adverse Event | 0 | 3 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Withdrawal of consent | 0 | 0 | 1
Not completed — Patients not treated | 2 | 3 | 1
Not completed — Not eligible for subsequent cycles | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population which included all randomized patients receiving the active study drug and HEC or MEC. Following the intent-to-treat principle, patients were assigned to the study treatment group according to the randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palonosetron 10 mcg/kg | Palonosetron 20 mcg/kg | Ondansetron | Total
Number analyzed (Participants) | 166 | 165 | 162 | 493
Age, Customized [Number; unit: participants]
  <2 years | 15 | 15 | 15 | 45
  2 to <6 years | 54 | 54 | 54 | 162
  6 to <12 years | 46 | 46 | 44 | 136
  12 to <17 years | 51 | 50 | 49 | 150
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 76 | 98 | 262
  Male | 78 | 89 | 64 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 26 | 12 | 64
  Not Hispanic or Latino | 140 | 139 | 150 | 429
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 0 | 2
  White | 156 | 154 | 159 | 469
  More than one race | 5 | 11 | 3 | 19
  Unknown or Not Reported | 1 | 0 | 0 | 1
Emetogenicity of chemotherapy in Cycle 1 [Number; unit: participants]
  MEC | 112 | 116 | 111 | 339
  HEC | 54 | 49 | 51 | 154

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Complete Response 0 to 24 Hours (Acute Phase) in Cycle 1
Description: Complete Response (CR) was defined as no vomiting, no retching, and no use of antiemetic rescue medication from 0 to 24 hours (acute phase) after T0 (start of administration of the most emetogenic chemotherapy) during first cycle. Time 0 (T0) is defined as the time when the patient starts the first cycle of chemotherapy.
Time Frame: 0 to 24 hours after T0
Population: Full Analysis Set (FAS) population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Palonosetron 10 mcg/kg | Palonosetron 20 mcg/kg | Ondansetron
Number analyzed (Participants) | 166 | 165 | 162
percentage of patients | 54.2 [46.3 to 61.9] | 59.4 [51.5 to 66.9] | 58.6 [50.6 to 66.2]
Statistical Analysis 1: Comparison: Palonosetron 20 mcg/kg vs Ondansetron; The stratum adjusted Mantel-Haenszel method was used to compute the confidence interval (CI) of the difference in proportion. If the lower bound of the 97.5% CI of either the difference (CR0-24h palonosetron 20 mcg/kg - CR0-24h ondansetron) or the difference (CR0-24h palonosetron 10 mcg/kg - CR0-24h ondansetron) was strictly superior to the non-inferiority margin (δ=-0.15) then the null hypothesis (H0) was rejected. A power of 80% was used for sample size computation; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 15% at an alpha level of 2.5% in a 1-sided test (equivalent to 5.0% 2-sided test) to reject the null hypothesis that the study drug was inferior to the active control drug by more than the non-inferiority margin; Risk Difference (RD) = 0.36, 97.5% CI 2-sided [-11.7 to 12.4]
Statistical Analysis 2: Comparison: Palonosetron 10 mcg/kg vs Ondansetron; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = -4.4, 97.5% CI 2-sided [-16.4 to 7.6]

2. Secondary Outcome: Proportion of Patients With Complete Response >24 to 120 Hours (Delayed Phase) in Cycle 1
Description: Complete Response (CR) was defined as no vomiting, no retching, and no use of antiemetic rescue medication from >24 to 120 hours (delayed phase) after T0 (start of administration of the most emetogenic chemotherapy) during first cycle.
Time Frame: from >24 to 120 hours (delayed phase) after T0
Population: Full Analysis Set (FAS) population.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Palonosetron 10 mcg/kg | Palonosetron 20 mcg/kg | Ondansetron
Number analyzed (Participants) | 166 | 165 | 162
percentage of patients | 28.9 [22.3 to 36.5] | 38.8 [31.4 to 46.7] | 28.4 [21.7 to 36.1]

ADVERSE EVENTS:
Description: Safety population (SAF), which allocated patients to treatment groups based on the treatment actually received. Patients received study treatment on Study Day 1 of each cycle for up to 4 cycles. The number of patients included in the SAF at each cycle was the following: 494 (cycle 1), 260 (cycle 2), 146 (cycle 3) and 69 (cycle 4).
Arm/Group | Palonosetron 10 mcg/kg | Palonosetron 20 mcg/kg | Ondansetron
Serious Adverse Events (participants affected / at risk) | 68/167 | 62/163 | 70/164
Other Adverse Events (participants affected / at risk) | 143/167 | 130/163 | 145/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palonosetron 10 mcg/kg (N=167) | Palonosetron 20 mcg/kg (N=163) | Ondansetron (N=164)
Febrile neutropenia (Blood and lymphatic system disorders) | 27 (31) | 30 (38) | 23 (35)
Anaemia (Blood and lymphatic system disorders) | 17 (21) | 14 (17) | 15 (17)
Neutropenia (Blood and lymphatic system disorders) | 12 (14) | 10 (13) | 11 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (17) | 8 (11) | 9 (11)
Leukopenia (Blood and lymphatic system disorders) | 10 (12) | 4 (7) | 9 (16)
Pancytopenia (Blood and lymphatic system disorders) | 6 (9) | 2 (2) | 6 (6)
Infection (Infections and infestations) | 4 (4) | 1 (1) | 3 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 3 (3) | 7 (7)
White blood cell count decreased (Investigations) | 6 (9) | 6 (8) | 4 (4)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Caecitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 3 (4) | 1 (1) | 2 (3)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 3 (3) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute disseminated encephalomyelitis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal tubular disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Aplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palonosetron 10 mcg/kg (N=167) | Palonosetron 20 mcg/kg (N=163) | Ondansetron (N=164)
Anaemia (Blood and lymphatic system disorders) | 65 (107) | 60 (89) | 61 (105)
Thrombocytopenia (Blood and lymphatic system disorders) | 35 (69) | 33 (61) | 37 (90)
Leukopenia (Blood and lymphatic system disorders) | 37 (74) | 27 (59) | 43 (104)
Neutropenia (Blood and lymphatic system disorders) | 35 (60) | 31 (51) | 22 (40)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (13) | 4 (4) | 4 (7)
Vomiting (Gastrointestinal disorders) | 13 (21) | 17 (39) | 22 (31)
Abdominal pain (Gastrointestinal disorders) | 15 (20) | 13 (16) | 18 (24)
Stomatitis (Gastrointestinal disorders) | 11 (15) | 12 (14) | 12 (16)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 6 (7) | 14 (15)
Constipation (Gastrointestinal disorders) | 8 (9) | 10 (12) | 8 (9)
Nausea (Gastrointestinal disorders) | 8 (10) | 6 (8) | 13 (19)
Pyrexia (General disorders) | 32 (40) | 19 (35) | 21 (38)
White blood cell count decreased (Investigations) | 12 (14) | 15 (18) | 15 (24)
Platelet count decreased (Investigations) | 10 (13) | 9 (12) | 10 (19)
Headache (Nervous system disorders) | 17 (24) | 9 (10) | 16 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 4 (4) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Sponsor does not submit a publication regarding the study to a journal within 12 months from study data analysis completion, the Investigator may publish an analysis of the study data collected as a result of the conduct of the study by the Investigator. The Investigator shall ensure that at least 60 days prior to submitting/presenting a manuscript/material relating to study to publishers a copy of all manuscripts/materials is provided to the Sponsor to allow the Sponsor sixty days to review.